CLINICAL TRIAL: NCT00404807
Title: Cardiac Function After CPAP Therapy in Patients With Chronic Heart Failure and Sleep Apnea. A Multicenter Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Sociedad Vasco-Navarra de Patología Respiratoria (Unknown); RESPIRA (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 01009
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Sleep Apnea; Heart Failure; Cardiovascular Diseases
Keywords: Continuous positive airway pressure; cardiovascular diseases; sleep apnea syndromes; sleep breathing disorders; sham CPAP
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure; Cardiovascular Diseases | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: CPAP(Continuous Positive Airway Pressure)

SUMMARY:
The role of continuous positive airway pressure (CPAP) in cardiac function in patients with CSA and OSA has been studied with varying results. Nevertheless, it is not clear whether CPAP treatment for respiratory sleep disorders in CHF could slow down deterioration or improve the cardiovascular function.

In an attempt to yield further insight into this subject, we undertook a multicentre study to analyze the role of CPAP therapy (optimal vs sham) in the LVEF and in other cardiac measurements in patients with CHF.Aim. We evaluated in a randomized multicentre placebo (sham-CPAP) controlled study the effect of CPAP treatment on the left ventricle ejection fraction (LVEF) among other cardiological related variables.

DETAILED DESCRIPTION:
From the Cardiologist Department of eight university hospitals CHF patients were referred to the Sleep Units with the sole condition of having a LVEF < 45%. After an interview and some clinical explorations, 127 out of 245 fulfilled the rigid inclusion and exclusion criteria in order to have CHF subjects without obvious comorbidity (see flowchart of figure 1). These subjects went to full (polysomnography) PSG. Fifty seven per cent of them (n: 73) had an apnea hypopnea index (AHI) > 10. Forty three per cent (n:54) had an AHI < 10. Only 17% of the patients had CSA. The selection and inclusion criteria used for recruitment were the following: 1) referral of patients with chronic heart failure to the sleep laboratory; 2) diagnosis of heart failure with at least one episode of cardiac failure; 3) LVEF less than 45% using radionuclide ventriculography; 4) clinical stability for at least one month prior to inclusion; 5) optimum treatment with diuretics and/or beta-blockers and/or digoxin and/or ACE inhibitors according to tolerance 6) no change in treatment for one month prior to inclusion; and 7) an Apnea-Hypopnea Index (AHI) greater than 10 measured by conventional polysomnography. The exclusion criteria were as follows: 1) patients that had a previous diagnosis of OSA or had been exposed to CPAP therapy. 2) uncontrolled arterial hypertension; 3) valvular or congenital cardiopathy, unstable angina, acute myocardial infarction or cardiac surgery in the three months prior to enrolment; 4) severe somnolence defined as severe sleepiness in situations of activity; 5) present or past medical history of clinically significant renal, liver or pulmonary disease; 6) untreated hypothyroidism; 7) clinically significant kyphoscoliosis; 8) morbid obesity with a body mass index (BMI)> 41 Kg/m2; and 9) concomitant use of the following drugs: morphine, hypnotics and sedatives, theophylline, acetazolamide or home oxygen therapy. Informed written consent was obtained from all subjects. This study was approved by the Human Ethics Committee of the 8 centres.

The subjects selected were randomized to receive CPAP or sham CPAP (Figure 1). They were evaluated at baseline (before any intervention) and after three months of follow-up. The assessment was performed on the basis of a LVEF. In addition, hypertension, subjective daytime sleepiness(sleepiness scale [ESS] (17), quality of life questionnaire according to the Spanish version of the SF-36 were also studied (18) The answers of the SF-36 were codified and divided into two groups, physical (PCS) and mental (MCS) with eight subclasses (physical function, physical role, bodily pain, general health, vitality, social function, emotional role, mental health). Other measurements were: dyspnea using the Borg scale (19), the New York Heart Association scale (NYHA scale), and the 6-minute walking test (20-21). The obstructive group accounting for 83% of all the patients were also studied. CPAP and sham CPAP compliance were recorded by a built-in device in the machine and registered at 4 weeks and at the end of the treatment period. After one month of treatment, another PSG was performed to re-assess the AHI. All visits were registered in a database on an encrypted website of the homepage of the Basque Health Service

ELIGIBILITY:
Inclusion Criteria:

1. referral of patients with chronic heart failure to the sleep laboratory;
2. diagnosis of heart failure with at least one episode of cardiac failure;
3. LVEF less than 45% using radionuclide ventriculography;
4. clinical stability for at least one month prior to inclusion;
5. optimum treatment with diuretics and/or beta-blockers and/or digoxin and/or ACE inhibitors according to tolerance
6. no change in treatment for one month prior to inclusion; and
7. an Apnea-Hypopnea Index (AHI) greater than 10 measured by conventional polysomnography

Exclusion Criteria:

1. patients that had a previous diagnosis of OSA or had been exposed to CPAP therapy.
2. uncontrolled arterial hypertension;
3. valvular or congenital cardiopathy, unstable angina, acute myocardial infarction or cardiac surgery in the three months prior to enrolment;
4. severe somnolence defined as severe sleepiness in situations of activity;
5. present or past medical history of clinically significant renal, liver or pulmonary disease;
6. untreated hypothyroidism;
7. clinically significant kyphoscoliosis;
8. morbid obesity with a body mass index (BMI)> 41 Kg/m2; and
9. concomitant use of the following drugs: morphine, hypnotics and sedatives, theophylline, acetazolamide or home oxygen therapy

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245
Dates: Start 2001-01; Study Completion 2004-06

PRIMARY OUTCOMES:
Ejection fraction

SECONDARY OUTCOMES:
Hypertension
Daytime sleepiness
Quality of life (SF-36)
NewYork Heart Scale (NYHA score),
Dyspnea (by using the Borg scale)
Exercise tolerance (6-min WT

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Egea-Santaolalla, MD, Principal Investigator — Hospital Universitario Txagorritxu. Vitoria Gasteiz. Spain
Locations (1):
- Hospital Universitario Txagorritxu, Vitoria-Gasteiz, Alava, Spain